CLINICAL TRIAL: NCT07259317
Title: A Phase 2, Single-Arm Trial of Relacorilant in Combination With Nab-Paclitaxel and Gemcitabine in Patients With Previously Untreated Metastatic Pancreatic Adenocarcinoma (TRIDENT)
Brief Title: Relacorilant With Nab-Paclitaxel and Gemcitabine in Patients With Metastatic Pancreatic Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CORT125134-558
Record Dates: First submitted 2025-11-03; First posted 2025-12-02 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Adenocarcinoma; Carcinoma, Pancreatic Ductal
Keywords: Pancreatic; Adenocarcinoma; PDAC; Pancreas
MeSH Terms: conditions — Adenocarcinoma; Carcinoma, Pancreatic Ductal | interventions — relacorilant; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Relacorilant in Combination with Nab-paclitaxel and Gemcitabine (Experimental): The patient will receive relacorilant 150 mg, administered orally under fed conditions, once daily for 3 consecutive days on the day before (excluding Cycle 1, day -1), the day of, and the day after nab-paclitaxel and gemcitabine infusions. Nab-paclitaxel (100 mg/m^2) and gemcitabine (1000 mg/m^2) will be administered by IV infusion on Days 1, 8, and 15 of each 28-day cycle. On days when relacorilant, nab-paclitaxel, and gemcitabine are administered, relacorilant will be administered first, then nab-paclitaxel, and gemcitabine last.
  Interventions: Drug: Relacorilant 150 mg once daily (QD); Drug: Nab-paclitaxel 100 mg/m^2; Drug: Gemcitabine 1000 mg/m^2

INTERVENTIONS:
Drug: Relacorilant 150 mg once daily (QD) — Relacorilant will be administered as capsules for oral dosing on the day before (excluding Cycle 1, Day -1), the day of, and the day after nab-paclitaxel and gemcitabine infusions.
  Other Names: CORT125134
Drug: Nab-paclitaxel 100 mg/m^2 — Nab-paclitaxel will be administered via intravenous (IV) infusion on Days 1, 8, and 15 of each 28-day cycle.
Drug: Gemcitabine 1000 mg/m^2 — Gemcitabine will be administered via intravenous (IV) infusion on Days 1, 8, and 15 of each 28-day cycle.

SUMMARY:
This is a Phase 2, single-arm study to evaluate the safety and efficacy of relacorilant in combination with nab-paclitaxel and gemcitabine in patients with previously untreated metastatic pancreatic adenocarcinoma (PDAC).

DETAILED DESCRIPTION:
Study treatment will be comprised of relacorilant, combined with nab-paclitaxel and gemcitabine. Each patient will receive relacorilant 150 mg administered orally under fed conditions, once daily for 3 consecutive days on the day before (excluding Cycle 1 Day -1), the day of, and the day after nab-paclitaxel (100 mg/m^2) and gemcitabine (1000 mg/m^2) infusions. Nab-paclitaxel and gemcitabine will be administered on Days 1, 8, and 15 of each 28-day cycle. Patients will receive study treatment until they reach progressive disease (PD), experience unmanageable toxicity, or until other discontinuation criteria are met.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form prior to screening procedures
* Histologic diagnosis or cytologic diagnosis of pancreatic adenocarcinoma (PDAC)
* Initial diagnosis of metastatic disease occurred ≤6 weeks prior to enrollment in the study
* Life expectancy of ≥3 months
* Radiographic confirmation of metastatic disease with at least 1 distant tumor metastasis measurable on radiology imaging per RECIST version 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Able to provide informed consent and comply with protocol requirements
* Able to swallow and retain oral medication and does not have uncontrolled emesis
* Has adequate gastrointestinal absorption
* Received no prior systemic anticancer therapy to treat metastatic disease
* If a patient received prior treatment of PDAC with chemotherapy, disease progression must have occurred >12 months after completing the last dose, and no persistent treatment-related toxicities can be present.
* Adequate organ function
* Negative pregnancy test for patients of childbearing potential
* Agree to use protocol defined precautions to avoid pregnancy

Exclusion Criteria:

* Any major surgery within 4 weeks prior to enrollment
* Prior treatment as follows:

  1. Radiotherapy, surgery, chemotherapy, immunotherapy, investigational therapy for the treatment of metastatic disease
  2. Systemic, inhaled, or prescription strength topical corticosteroids within 5 times the half-life of the corticosteroid used prior to first dose of study drug
* Received gemcitabine or nab-paclitaxel to treat their PDAC
* Known germline or somatic breast cancer gene (BRCA) mutation
* Peripheral neuropathy from any cause >Grade 1
* Medical conditions requiring chronic or frequent treatment with corticosteroids
* History of severe hypersensitivity or severe reaction to any of study drugs or their excipients
* Concurrent treatment with mifepristone or other glucocorticoid receptor modulators.
* Uncontrolled condition(s) which, may confound the results of the trial or interfere with the patient's safety or participation
* Active infection with HIV, hepatitis C or hepatitis B virus
* Known untreated parenchymal brain metastasis or uncontrolled central nervous system metastases
* History of other malignancy within 3 years prior to enrollment
* Taking protocol-prohibited medications
* Concurrent treatment with other investigational treatment studies for cancer
* Has received a live vaccine within 30 days prior to the study start date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 12 months
  To evaluate PFS as the time from enrollment until first documented progressive disease (PD) by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as determined by the Investigator, or death due to any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of enrollment until the date of death from any cause, whichever comes first, assessed up to 19 months
Best Overall Response (BOR) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 12 months
Objective Response Rate (ORR) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 12 months
  To evaluate the proportion of patients with measurable disease at Baseline who attain complete response (CR) or partial response (PR) by RECIST version 1.1.
Duration of Response (DoR) | From date of first objective response until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 12 months
  To evaluate DOR as the time from the first CR or PR to first documented PD or death, whichever comes first.
Clinical Benefit Rate (CBR) | Week 24
  To evaluate clinical benefit rate as the proportion of patients who attain CR, PR, or stable disease (SD) at Week 24 as per RECIST version 1.1.
Cancer Antigen 19-9 (CA19-9) Kinetics | Baseline to Weeks 4, 8, and 16
  To evaluate change in CA19-9 from baseline in patients who had an elevated baseline CA19-9 and change in CA19-9 at Weeks 4, 8, and 16 from baseline in all patients.
Number of Patients with 1 or More Adverse Events | Time of first dose up to 30 days after last dose
Maximum Plasma Concentration (Cmax) of Relacorilant | Pre- and postdose on Cycle 1 Day 8 (each cycle is 28 days)
Area Under the Plasma Concentration-time Curve (AUC) of Relacorilant | Pre- and postdose on Cycle 1 Day 8 (each cycle is 28 days)
Cmax of Nab-paclitaxel | Postdose on Cycle 1 Day 8 (each cycle is 28 days)
AUC of Nab-paclitaxel | Postdose on Cycle 1 Day 8 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Pai, Study Director — Corcept Therapeutics
Locations (1):
- Site 01, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No